

SEDE LEGALE: Corso Mazzini, 18 28100 Novara - Tel. 0321.3731 www.maggioreosp.novara.it

Cod. Fiscale - Part. IVA: 01521330033

## TITLE: Evaluation of the efficacy of the treatment of benign prostatic hypertrophy with Serenoa Repens extracted with CO2 + PEA (Palmitoylethanolamide) in monotherapy or in combination with tamsulosin. ProSeRePEA trial.

Novara, 02/17/2021



SEDE LEGALE: Corso Mazzini, 18 28100 Novara - Tel. 0321.3731 www.maggioreosp.novara.it

Cod. Fiscale - Part. IVA: 01521330033

## **Informed Consent – Participation in the study**

TITLE: Evaluation of the efficacy of the treatment of benign prostatic hypertrophy with Serenoa Repens extracted with CO2 + PEA (Palmitoylethanolamide) in monotherapy or in combination with tamsulosin. ProSeRePEA trial.

| PROMOTER: | |
|---|---|
| $\label{eq:continuous} \mbox{Dr Michele Billia, S.C.D.U. of Urology, A.O.U. Major of the}$ | Charity of Novara |
| COLLABORATORS: | |
| Prof. Alessandro Volpe, Dr. Silvia Cavalli, S.C.D.U. of Urology, A.O.U. Major of the Charity of Novara | |
| The undersigned | born on |
| (Name and Surname) | (Date of birth) |
| After having read the Information, he declares the following: | |
| • that I have read and understood the Information Sheet for | r the aforementioned study and that I have had ample time |
| and opportunity to ask questions and obtain satisfactory answ | ers from the investigator; |
| • that you understand that participation is voluntary and that you can withdraw from the study at any time, without | |
| having to give an explanation and without influencing your future medical care in any way; | |
| • to have understood that parts of his file, which show part | icipation in clinical research, may be viewed by the |
| Regulatory Authorities, the Ethics Committee and the Local Health Administration and, therefore, agrees that these | |
| subjects have access to his data. | |
| As a result of his statements: | |
| □ Accepts □ DOES NOT agree to freely participate in the afor | rementioned study. |
| $\square$ Accepts $\square$ DOES NOT agree to inform your GP regarding participation in this study. | |
| Date | |
| Investigator doctor | |
| (Name and surname) | |
| Date Investigator's signature | |

NOTES: 1 photocopy for the patient and the original to be kept in the patient's medical record